CLINICAL TRIAL: NCT03742349
Title: A Phase Ib, Multicenter, Open-label Dose Escalation and Expansion Platform Study of Select Immunotherapy Combinations in Adult Patients With Triple-negative Breast Cancer
Brief Title: Study of Safety and Efficacy of Novel Immunotherapy Combinations in Patients With Triple Negative Breast Cancer (TNBC).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a sponsor decision and was not a consequence of any safety concern
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CADPT01A12101C; 2018-002244-82 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: Phase Ib, TNBC, advanced, metastatic, immunotherapy, PDR001,; LAG525, NIR178, INC280, MCS110, ACZ885
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — spartalizumab; capmatinib; canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1: spartalizumab + LAG525 + NIR178 (Experimental): phase Ib (escalation and expansion)
  Interventions: Biological: spartalizumab; Biological: LAG525; Drug: NIR178
- 2: spartalizumab +LAG525 +capmatinib (Experimental): phase Ib (escalation and expansion)
  Interventions: Biological: spartalizumab; Biological: LAG525; Drug: capmatinib
- 3: spartalizumab + LAG525 + MCS110 (Experimental): phase Ib (escalation and expansion)
  Interventions: Biological: spartalizumab; Biological: LAG525; Biological: MCS110
- 4: spartalizumab +LAG525 +canakinumab (Experimental): phase Ib (escalation and expansion)
  Interventions: Biological: spartalizumab; Biological: LAG525; Biological: canakinumab

INTERVENTIONS:
Biological: spartalizumab — LIVI (Liquid in vial) Concentrate for Solution for infusion
  Other Names: PDR001
Biological: LAG525 — LAG525 LIVI (Liquid in vial) Concentrate for Solution for infusion
Drug: NIR178 — Capsule
  Arms: 1: spartalizumab + LAG525 + NIR178
Drug: capmatinib — Tablet
  Other Names: INC280
  Arms: 2: spartalizumab +LAG525 +capmatinib
Biological: MCS110 — LIVI (Liquid in vial) Concentrate for Solution for infusion
  Arms: 3: spartalizumab + LAG525 + MCS110
Biological: canakinumab — LIVI (Liquid in vial) Solution for injection
  Other Names: ACZ885
  Arms: 4: spartalizumab +LAG525 +canakinumab

SUMMARY:
This is a Phase Ib, open label, dose escalation study of spartalizumab + LAG525 in combination with NIR178, capmatinib, MCS110, or canakinumab, followed by a dose expansion in adult patients with advanced or metastatic TNBC.

During the dose-escalation part of each treatment arm, patients will be treated with fixed doses of spartalizumab + LAG525 in combination with partner investigational drugs to be escalated until the MTD is reached or a lower RDE is established: NIR178, capmatinib, MCS110, or canakinumab. It is anticipated that other partner study drugs may be added in the future by protocol amendment.

After the determination of the MTD/RDE for a particular treatment arm, dose expansion may begin in that arm in order to further assess safety, tolerability, PK/PD, and anti-tumor activity of each combination at the MTD/RDE. Dose expansion arms may initiate only after consideration by the Investigators and Novartis of all available toxicity information, the assessment of risk to future patients from the BLRM, and the available PK, preliminary efficacy, and PD information. There is no requirement for dose-escalation treatment arms reaching an MTD/RDE to proceed to dose expansion.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with advanced/metastatic TNBC (defined as HER-2 negative with <1% of tumor cell nuclei immunoreactive for estrogen receptor (ER) and progesterone receptor (PR)), with measurable disease as determined by RECIST version 1.1 (refer to Appendix 16.1). Tumor lesions previously irradiated or subjected to other loco-regional therapy will only be considered measurable if there is documented disease progression at the treated site prior to study entry.
* Patients should have received standard chemotherapy for advanced or metastatic disease but should not have received more than 2 prior lines of chemotherapy. Neoadjuvant or adjuvant chemotherapy will count as one prior line.
* Patients must have received prior systemic treatment that included taxane-based chemotherapy for neoadjuvant or metastatic disease.
* Patients must have a site of disease amenable to core needle biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patients must be willing to undergo a new tumor biopsy at screening, and during therapy on the study. Exceptions may be considered after documented discussion with Novartis. Patients with available archival tumor tissue obtained ≤6 months prior to study treatment initiation do not need to undergo a new tumor biopsy at screening, if the patient has not received any anti-cancer therapy since the biopsy was taken, and if adequate tissue is available.

Main exclusion criteria applicable to all treatment arms:

* Patient has received prior treatment with anti-LAG-3, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody (any line of therapy).
* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within 2 weeks prior to initiating study treatment.
* History of severe hypersensitivity reactions to any ingredient of study drug(s) and other mAbs and/or their excipients.
* Impaired cardiac function or clinically significant cardiac disease.
* HIV infection.
* Patients with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, including those with inactive disease for patients receiving either capmatinib, MCS110 or canakinumab.
* Active, known or suspected autoimmune disease.
* History of or current interstitial lung disease or pneumonitis grade ≥ 2.
* Subjects with tuberculosis (TB), for patients receiving either MCS110 or canakinumab.

Other eligibility criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | at month 18
  Month 18 is assumed to be study end
Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of safety | at month 18
  Month 18 is assumed to be study end
Incidence of dose limiting toxicities (DLTs) of treatment (Escalation only) | at Day 28
  end of first cycle
Frequency of dose interuptions | at month 18
  Month 18 is assumed to be study end
Frequency of dose reductions | at month 18
  Month 18 is assumed to be study end
Dose intensities | at month 18
  Month 18 is assumed to be study end

SECONDARY OUTCOMES:
Best overall response (BOR) | at month 18
  Month 18 is assumed to be study end
Progression free survival (PFS) per RECIST v1.1 and iRECIST | at month 18
  Month 18 is assumed to be study end
Presence of anti-spartalizumab antibodies | at Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
Presence of anti-LAG525 antibodies | at Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
Presence of anti-MCS110 antibodies | at Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
Presence of anti-canakinumab antibodies | at Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
Serum concentration of spartalizumab, LAG525, MCS110, canakinumab | at Day 1, Day 8, Day 15, Day 29, Day 57, Day 65, Day 70, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
Plasma concentration of NIR178, NJI675, capmatinib | at Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 197, Day 253, Day 309 and EOT
PK parameter (Tmax) of spartalizumab | at month 12
  cycle 12
PK parameter (Cmax) of spartalizumab | at month 12
  cycle 12
PK parameter (AUC) of spartalizumab | at month 12
  cycle 12
PK parameter (Tmax) of LAG525 | at month 12
  cycle 12
PK parameter (Cmax) of LAG525 | at month 12
  cycle 12
PK parameter (AUC) of LAG525 | at month 12
  cycle 12
PK parameter (Tmax) of NIR178 | at month 12
  cycle 12
PK parameter (Cmax) of NIR178 | at month 12
  cycle 12
PK parameter (AUC) of NIR178 | at month 12
  cycle 12
PK parameter (Tmax) of capmatinib | at month 12
  cycle 12
PK parameter (Cmax) of capmatinib | at month 12
  cycle 12
PK parameter (AUC) of capmatinib | at month 12
  cycle 12
PK parameter (Tmax) of MCS110 | at month 12
  cycle 12
PK parameter (Cmax) of MCS110 | at month 12
  cycle 12
PK parameter (AUC) of MCS110 | at month 12
  cycle 12
PK parameter (Tmax) of canakinumab | at month 12
  cycle 12
PK parameter (Cmax) of canakinumab | at month 12
  cycle 12
PK parameter (AUC) of canakinumab | at month 12
  cycle 12
Changes from baseline of PD markers in tumor tissue (TILs, CD8, PD-L1, LAG-3) | at baseline and at Day 43

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Columbia University Medical Center- New York Presbyterian Columbia, New York, New York
  - Sarah Cannon Research Institute Sarah Cannon Research, Nashville, Tennessee
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Novartis Investigative Site, Shatin, New Territories, Hong Kong, Hong Kong
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18138
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2282